CLINICAL TRIAL: NCT02070354
Title: Physical Fitness and Macro- and Micro- Nutrient Intake in a Morbidly Obese Bariatric Surgery Population
Brief Title: Physical Fitness and Nutrition Intake in Bariatric Surgery Population
Status: Completed | Type: Observational
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0182
Record Dates: First submitted 2014-02-19; First posted 2014-02-25 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Physical Activity; Nutrition; Weight Loss
MeSH Terms: conditions — Obesity; Motor Activity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Group 1: New clinic visit in GI Nutrition (prior to bariatric surgery).
- Group 2: 1 month prior to bariatric surgery
- Group 3: 6 months after bariatric surgery
- Group 4: 12 months after bariatric surgery
- Group 5: 24 months after bariatric surgery
- Group 6: ≥ 36 months after bariatric surgery

SUMMARY:
The purpose of this research study is to determine how bariatric surgery affects physical activity and nutrient intake.

This research study is being done because the investigators want to determine better recommendations to provide to bariatric surgery patients.

DETAILED DESCRIPTION:
This is a two-pronged study. The first phase is a cross-sectional study design meaning each participant will only be tested once. The investigators wish to test patients from each of the groups listed below to determine CR fitness, activity level, and nutrient intake. The investigators wish to determine if any improvements from bariatric surgery can be maintained over a 2-year period following surgery. If this is the case, our next project will be to track the patients recruited at their new visit longitudinally at all of the five time points listed below.

1. New visit with GI Nutrition
2. 1 month prior to bariatric surgery (at the time of the patient's initial visit with the surgeon (6-7 months after their new visit))
3. 6 months after bariatric surgery
4. 12 months after bariatric surgery
5. 24 months after bariatric surgery

ELIGIBILITY:
Inclusion Criteria:

* Competent patients enrolled in the pre- or post-operative bariatric surgery program at the Center for Nutrition and Weight Management at GMC, Danville, PA.
* Ability to perform a 6 Minute Walk Test.
* Aged 18 through 70.
* Willingness to receive dietary recall phone calls and accessibility to a telephone.

Exclusion Criteria:

* Patients with severe lung disease requiring oxygen therapy.
* Pulmonary embolus or pulmonary infarction.
* Patients with cardiopulmonary disease (e.g., prior myocardial infarction, coronary artery bypass, or vascular stent).
* Unstable angina.
* Uncontrolled cardiac dysrhythmias causing symptoms or hemodynamic compromise.
* Patients with any health reason that limits walking.
* Patients with a temporary injury that limits walking.
* Patients who use a wheelchair, other assistive device for walking, or have difficulty ambulating during activities of daily living.
* Patients predetermined to be illiterate or incompetent.
* Patients who are currently pregnant or have been pregnant at any time since bariatric surgery.
* Tobacco use.
* Patients with electronic defibrillators or other embedded electronic medical devices.
* Acute systemic infection, accompanied by fever, body aches, or swollen lymph glands
* Patients who have undergone revisional bariatric surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 210 Geisinger subjects will participate in this study. Participants will be volunteers from the patient population of the Center for Nutrition and Weight Management between the ages of 18 and 70 years.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2009-08; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pre-Operative 6 Min Walk Test | Pre-operative
  6 Min Walk for Distance
1 Month Post-Operative 6 Min Walk Test | 1 Month Post-Operative
  6 Min Walk for Distance
6 Month Post-Operative 6 Min Walk Test | 6 Month Post-Operative
  6 Min Walk for Distance
12 Month Post-Operative 6 Min Walk Test | 12 Month Post-Operative
  6 Min Walk for Distance
24 Month Post-Operative 6 Min Walk Test | 24 Month Post-Operative
  6 Min Walk for Distance
Peak Oxygen Uptake (peak VO2) | 36 Month Post-Operative
  Measured using an incremental exercise test on an electronically breaked bike and indirect calorimetry.

SECONDARY OUTCOMES:
Pre-operatively Physical activity | Pre-operatively
  Measured using 7 days of accelerometry (actigraph).
1 Month Post-Operative Physical activity | 1 Month Post-Operative
  Measured using 7 days of accelerometry (actigraph).
6 Month Post-Operative Physical activity | 6 Month Post-Operative
  Measured using 7 days of accelerometry (actigraph).
12 Month Post-Operative Physical activity | 12 Month Post-Operative
  Measured using 7 days of accelerometry (actigraph).
24 Month Post-Operative Physical activity | 24 Month Post-Operative
  Measured using 7 days of accelerometry (actigraph).
36 Month Post-Operative Physical activity | 36 Month Post-Operative
  Measured using 7 days of accelerometry (actigraph).

OTHER OUTCOMES:
Pre-operative Dietary Intake | Pre-operatively
  Measured using three 24 h dietary recalls.
1 Month Post-operative Dietary Intake | 1 Month Post-operative
  Measured using three 24 h dietary recalls.
12 Month Post-operative Dietary Intake | 12 Month Post-operative
  Measured using three 24 h dietary recalls.
24 Month Post-operative Dietary Intake | 24 Month Post-operative
  Measured using three 24 h dietary recalls.
Post-operative Dietary Intake | 36 Month Post-operative
  Measured using three 24 h dietary recalls.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D. Still, DO, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States